CLINICAL TRIAL: NCT02933814
Title: Liposomal Bupivacaine in Ambulatory Hand Surgery
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Inadequate number of subjects meet study criteria
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Subhas Gupta, MD, PhD, Chair of the Department of Plastic Surgery, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5150445
Record Dates: First submitted 2016-10-04; First posted 2016-10-14 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients in Group 1 (Plain Bupivacaine) will be treated intra-operatively with injections of 0.25% bupivacaine, with 10 mL (25 mg) delivered to perform a field block of the soft tissue and subfascial plane at the initiation of the surgical procedure.
- Experimental Group (Experimental): Patients in Group 2 (Liposomal Bupivacaine + Plain Bupivacaine) will be treated intra-operatively with the initial injection of 0.25% bupivacaine 5 - 10 mL (12.5 - 25 mg) delivered to perform a field block of the soft tissue and subfascial plane at the initiation of the procedure.
  Interventions: Drug: Liposomal Bupivicaine

INTERVENTIONS:
Drug: Liposomal Bupivicaine — Patients in Group 2 (Liposomal Bupivacaine + Plain Bupivacaine) will be treated intra-operatively with the initial injection of 0.25% bupivacaine 5 - 10 mL (12.5 - 25 mg) delivered to perform a field block of the soft tissue and subfascial plane at the initiation of the procedure.
  Other Names: Exparel
  Arms: Experimental Group

SUMMARY:
This study is being done to evaluate pain management regimens following ambulatory hand surgery. Improved pain control may be associated with decreased complications, decreased pain scores, decreased opioid dependence, improved patient comfort and satisfaction, and reduced healthcare costs. Liposomal bupivacaine is an FDA-approved local anesthetic. There will be two groups. One group will receive liposomal bupivacaine. One group will not. The results will be compared.

Patients will be over the age of 18 ambulatory hand surgery. Approximately 40 subjects will participate in this study at LLU.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and over undergoing ambulatory hand surgery involving soft tissue and subfascial structures, including: CMC arthritis, flexor and extensor tendon injury, symptomatic ganglia, hand and finger fractures

Exclusion Criteria:

* Patients who are unable to give informed consent to participate in this study
* Patients with a documented history of hypersensitivity reactions to local anesthetic agents
* Patients with a diagnosis of chronic pain disorders such as fibromyalgia, chronic migraine headaches, or psychiatric disorders other than depression or anxiety
* Patients who are currently pregnant
* Patients with impaired hepatic function
* Patients with underlying nerve damage or impairment
* Patients with renal impairment/failure
* Patients whose career/livelihood require a great deal of hand dexterity, in whom a complication could cause a significant impact on life and career (ex: musician, dentist)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-09 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Post-operative Opioid Use | At scheduled intervals up to 168 hours post-operatively
  Patients will record their opioid use post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Subhas Gupta, MD, Principal Investigator — Chair of the Department of Plastic Surgery
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No